CLINICAL TRIAL: NCT07141381
Title: A Phase 1, Open-label, 3-Period, Randomized 2-Sequence Study to Evaluate the Effect of Food and a Proton Pump Inhibitor on the Pharmacokinetics of VRN110755 in Healthy Adult Participants
Brief Title: A Study to Evaluate the Effect of Food and a Proton Pump Inhibitor on the Pharmacokinetics of VRN110755
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Voronoi, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VRN110755-001
Record Dates: First submitted 2025-07-24; First posted 2025-08-26 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Fasted → Fed → Fed with PPI (Experimental): Participants in this sequence will receive VRN110755 80 mg orally under the following conditions across three periods:
  Period 1: Fasted state Period 2: Fed state (standard high-fat meal) Period 3: Fed state after 5 days of rabeprazole 20 mg daily
  Interventions: Drug: VRN110755
- Sequence 2: Fed → Fasted → Fasted with PPI (Experimental): Participants in this sequence will receive VRN110755 80 mg orally under the following conditions across three periods:
  Period 1: Fed state (standard high-fat meal) Period 2: Fasted state Period 3: Fasted state after 5 days of rabeprazole 20 mg daily
  Interventions: Drug: Rabeprazole

INTERVENTIONS:
Drug: VRN110755 — VRN110755 is an investigational EGFR inhibitor administered as an 80 mg oral capsule. It will be given to all participants under fasted, fed, and PPI pre-treated conditions across three periods in a crossover design.
  Arms: Sequence 1: Fasted → Fed → Fed with PPI
Drug: Rabeprazole — Rabeprazole 20 mg will be administered orally once daily for 5 days prior to VRN110755 dosing in Period 3. This is to assess the effect of increased gastric pH (via proton pump inhibition) on the pharmacokinetics of VRN110755.
  Arms: Sequence 2: Fed → Fasted → Fasted with PPI

SUMMARY:
This is a Phase 1, open-label, randomized, single-center study to evaluate the effect of food and a proton pump inhibitor (PPI) on the pharmacokinetics (PK) of VRN110755 in healthy adult participants. The primary aim of this study is to assess the impact of food and rabeprazole co-administration on the systemic exposure of VRN110755. Safety and tolerability will also be evaluated.

DETAILED DESCRIPTION:
The study consists of two treatment sequences in a 3-period, crossover design. Approximately 24 healthy adult participants will be randomized 1:1 to one of the following sequences:

Sequence 1: Participants will receive VRN110755 80 mg orally in the fasted state (Period 1), then in the fed state (Period 2), and finally in the fed state with 5 days of rabeprazole pre-treatment (Period 3).

Sequence 2: Participants will receive VRN110755 80 mg orally in the fed state (Period 1), then in the fasted state (Period 2), and finally in the fasted state with 5 days of rabeprazole pre-treatment (Period 3).

Rabeprazole 20 mg will be administered orally once daily for 5 consecutive days prior to the final dosing of VRN110755 in Period 3.

All participants will remain under clinical observation for safety monitoring and pharmacokinetic sampling throughout each period. Blood and urine samples will be collected at defined intervals for the analysis of VRN110755 and its metabolites.

Each participant's total study duration will be approximately 76 days, including screening, treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged between 18 and 65 years, inclusive, at the time of informed consent.
2. In good general health, with no significant medical history and no clinically significant abnormalities on physical examination, as determined by the investigator.
3. Body mass index (BMI) between 18.0 and 32.0 kg/m², and weight ≥ 50 kg at screening.
4. Clinical laboratory values within normal ranges, unless deemed not clinically significant by the investigator.
5. Female participants of childbearing potential who are sexually active with a male partner must agree to use highly effective contraception methods from screening through 6 months after the last dose of investigational product.
6. Female participants must have a negative pregnancy test at screening and pre-dose.
7. Women not of childbearing potential must be surgically sterile or postmenopausal for ≥12 months.
8. Male participants must agree to use barrier contraception in conjunction with a highly effective method if engaging with women of childbearing potential, from screening through 6 months after the last dose.
9. Male participants must not donate sperm, and female participants must not donate ova, from the first dose through 6 months after the last dose.
10. Able and willing to comply with study procedures and site visits.
11. Able and willing to provide written informed consent before any study procedures are performed.

Exclusion Criteria:

1. Any significant medical or psychiatric condition that may interfere with study participation or interpretation of results, as determined by the investigator.
2. Clinically significant abnormal ECG findings, including QTcF > 450 ms (males) or > 470 ms (females).
3. Abnormal vital signs at screening (e.g., systolic BP > 140 or < 90 mmHg, diastolic BP > 90 or < 60 mmHg, or history of symptomatic hypotension).
4. Active liver disease, or AST/ALT > 1.5 × upper limit of normal.
5. Known or suspected gastrointestinal disorders that may interfere with drug absorption (e.g., IBD, chronic diarrhea, malabsorption).
6. Positive urine drug screen or alcohol breath test at screening.
7. Regular alcohol use >14 standard drinks/week or >3 drinks/day.
8. Positive test for HIV, Hepatitis B (HBsAg), or Hepatitis C antibody.
9. History of severe allergies or anaphylaxis, or known hypersensitivity to study drug components.
10. Recent infections requiring parenteral antibiotics within 6 months before first dose.
11. Vaccination with live vaccine within 4 weeks prior to first dose.
12. Blood donation >400 mL within 60 days, or component donation within 30 days prior to dosing.
13. eGFR ≤ 90 mL/min/1.73 m² at screening.
14. Use of nicotine-containing products within 7 days before dosing or unwillingness to abstain during the study.
15. Use of prescription/OTC medications, herbal products, or supplements within 14 days prior to dosing, unless approved by the investigator.
16. Use of CYP3A4 inhibitors/inducers or medications affecting metabolism of VRN110755 within 14 days prior to dosing.
17. Unwillingness to follow dietary restrictions (e.g., cannot consume high-fat meals).
18. Use of proton pump inhibitors, H2 blockers, or antacids within 8 weeks prior to first dose (except planned rabeprazole use in study).
19. Known hypersensitivity to PPIs (e.g., rabeprazole).
20. Planned or current participation in another investigational trial or use of another investigational product within 30 days or 5 half-lives.
21. Poor peripheral venous access.
22. Any condition that, in the opinion of the investigator, would jeopardize participant safety or interfere with study compliance or data integrity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2025-12-17 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUC₀-inf) of VRN110755 | Up to 312 hours post-dose (for each treatment period)
  To evaluate the effect of food and rabeprazole on the extent of systemic exposure of VRN110755 by measuring AUC₀-inf under fasted, fed, and PPI conditions.
Maximum Observed Plasma Concentration (Cmax) of VRN110755 | Up to 312 hours post-dose (for each treatment period)
  To assess the peak plasma concentration of VRN110755 under different dosing conditions (fasted, fed, fed/fasted + PPI).
Time to Maximum Observed Concentration (Tmax) of VRN110755 | Up to 312 hours post-dose (for each treatment period)
  To assess the time to reach peak concentration of VRN110755 after single-dose oral administration under different conditions.
Comparison of Pharmacokinetic Parameters (AUC and Cmax Ratios) Across Treatment Conditions | Up to 312 hours post-dose (for each treatment period)
  To compare AUC and Cmax values of VRN110755 between fed vs. fasted, and PPI vs. non-PPI conditions using statistical analysis.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From Day 1 of Period 1 through the End of Study (approximately 76 days per participant)
  To evaluate the safety and tolerability of single oral doses of VRN110755 administered under fasted, fed, and PPI conditions by assessing the incidence, severity, and relationship of TEAEs.
Incidence of Serious Adverse Events (SAEs) | From Day 1 of Period 1 through the End of Study (approximately 76 days per participant)
  To monitor and document any SAEs occurring after VRN110755 administration under any treatment condition.
Number of Participants with Abnormal Clinical Laboratory Test Results | Baseline (Day 1), pre-dose on Day 15 and Day 34, and End-of-Study Visit (Day 48)
  The number of participants exhibiting abnormal laboratory values in hematology, biochemistry, coagulation, or urinalysis assessments..
Change in 12-lead ECG Parameters From Baseline | Baseline (Day 1), pre-dose on Day 15 and Day 34, and End-of-Study Visit (Day 48)
  Change from baseline in ECG parameters, including heart rate, PR interval, QRS duration, QT interval, and QTcF (Fridericia). ECGs will be recorded after at least 5 minutes of rest in the supine position. Triplicate ECGs will be taken at screening; single ECGs will be performed at other scheduled timepoints unless clinically indicated.
Change in Systolic Blood Pressure From Baseline | Baseline (Day 1), pre-dose on Day 15 and Day 34, and End-of-Study Visit (Day 48).
  Change from baseline in systolic blood pressure measured after at least 5 minutes of rest in the supine position. Triplicate readings will be performed at pre-dose; single measurements at other scheduled timepoints.
Change in Diastolic Blood Pressure From Baseline | Baseline (Day 1), pre-dose on Day 15 and Day 34, and End-of-Study Visit (Day 48).
  Change from baseline in diastolic blood pressure measured after at least 5 minutes of rest in the supine position. Triplicate readings will be performed at pre-dose; single measurements at other scheduled timepoints.
Change in Pulse Rate From Baseline | Baseline (Day 1), pre-dose on Day 15 and Day 34, and End-of-Study Visit (Day 48).
  Change from baseline in pulse rate measured after at least 5 minutes of rest in the supine position. Triplicate readings will be performed at pre-dose; single measurements at other scheduled timepoints.
Change in Respiratory Rate From Baseline | Baseline (Day 1), pre-dose on Day 15 and Day 34, and End-of-Study Visit (Day 48).
  Change from baseline in respiratory rate measured after at least 5 minutes of rest in the supine position. Triplicate readings will be performed at pre-dose; single measurements at other scheduled timepoints.
Change in Tympanic Temperature From Baseline | Baseline (Day 1), pre-dose on Day 15 and Day 34, and End-of-Study Visit (Day 48).
  Change from baseline in tympanic temperature measured after at least 5 minutes of rest in the supine position. Triplicate readings will be performed at pre-dose; single measurements at other scheduled timepoints.
Cumulative Amount Excreted (Ae) of VRN110755 | 0 to 24 hours post-dose in each study period.
  Cumulative amount of VRN110755 excreted in urine, measured over 0 to 24 hours post-dose under different study conditions.
Fraction Excreted (Fe) of VRN110755 | 0 to 24 hours post-dose in each study period.
  Fraction of the administered dose of VRN110755 excreted in urine, measured over 0 to 24 hours post-dose under different study conditions.
Renal Clearance (CLr) of VRN110755 | 0 to 24 hours post-dose in each study period.
  Renal clearance of VRN110755, determined from urinary excretion and plasma concentration data under different study conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No